CLINICAL TRIAL: NCT01341652
Title: Randomized Phase II Trial of a DNA Vaccine Encoding Prostatic Acid Phosphatase (pTVG-HP) Versus GM-CSF Adjuvant in Patients With Non-Metastatic Prostate Cancer
Brief Title: Phase II PAP Plus GM-CSF Versus GM-CSF Alone for Non-metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO08801; 2013-1679 (Other: Institutional Review Board); NCI-2011-00965 (Registry Identifier: NCI CTRP); A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison); Protocol Version 10/7/2015 (Other: UW Madison)
Record Dates: First submitted 2011-03-24; First posted 2011-04-26 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — regramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- pTVG-HP vaccine with GM-CSF (Experimental): pTVG-HP (100 µg) with rhGM-CSF (208 µg) administered intradermally (i.d.) biweekly for 6 total doses, then every 3 months to complete a 2-year treatment period
  Interventions: Biological: pTVG-HP
- GM-CSF alone (Active Comparator): rhGM-CSF (208 µg) administered intradermally (i.d.) biweekly for 6 total doses, then every 3 months to complete a 2-year treatment period
  Interventions: Biological: rhGM-CSF

INTERVENTIONS:
Biological: pTVG-HP — pTVG-HP (100 µg) with rhGM-CSF (208 µg) administered intradermally (i.d.) biweekly for 6 total doses, then every 3 months to complete a 2-year treatment period
  Arms: pTVG-HP vaccine with GM-CSF
Biological: rhGM-CSF — rhGM-CSF (208 µg) administered intradermally (i.d.) biweekly for 6 total doses, then every 3 months to complete a 2-year treatment period
  Other Names: GM-CSF; granulocyte-macrophage colony-stimulating factor
  Arms: GM-CSF alone

SUMMARY:
The investigators are trying to find new methods to treat prostate cancer. The approach the investigators are taking is to try to enhance patients' own immune response against the cancer. In this study the investigators will be testing the effectiveness of a vaccine that may be able to help the body fight prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of adenocarcinoma of the prostate
* Completion of local therapy by surgery and/or ablative radiation therapy at least 3 months prior to entry, with removal or ablation of all visible disease, including seminal vesical and/or local lymph node involvement
* Rising prostate specific antigen (PSA) levels without scan evidence of metastatic disease
* Asymptomatic or mildly symptomatic and life expectancy of at least 4 months

Exclusion Criteria:

* Small cell or other variant prostate cancer histology
* Evidence of immunosuppression
* Prior treatment with androgen deprivation except if given neoadjuvantly or adjuvantly with radiation therapy or at time of prostatectomy. In this situation, no more than 24 months of androgen deprivation must have been given and treatment must not have been within 12 months prior to screening for this study.
* Serum testosterone at screening < 50 ng/dL
* Known bone metastases or lymph node involvement as determined by bone scan or computed tomography (CT) scan of the abdomen and pelvis within 4 weeks of study entry
* Prior vaccine therapy for prostate cancer
* Known allergic reactions to granulocyte-macrophage colony-stimulating factor (GM-CSF)
* Severe intercurrent medical conditions or laboratory abnormalities that would impart, in the judgment of the Medical Monitor, excess risk associated with study participation or study agent administration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-05-23 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, M.D., PhD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] McNeel DG, Eickhoff JC, Johnson LE, Roth AR, Perk TG, Fong L, Antonarakis ES, Wargowski E, Jeraj R, Liu G. Phase II Trial of a DNA Vaccine Encoding Prostatic Acid Phosphatase (pTVG-HP [MVI-816]) in Patients With Progressive, Nonmetastatic, Castration-Sensitive Prostate Cancer. J Clin Oncol. 2019 Dec 20;37(36):3507-3517. doi: 10.1200/JCO.19.01701. Epub 2019 Oct 23. PMID 31644357
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety-nine participants were enrolled between 2011 and 2016 at the University of Wisconsin; University of California, San Francisco; and Johns Hopkins University.
Period: Overall Study
Arm/Group | GM-CSF Alone | pTVG-HP Vaccine With GM-CSF
Started | 49 | 50
Completed | 49 | 48
Not Completed | 0 | 2
Not completed — Incorrect Random Assignment | 0 | 1
Not completed — ineligible; presence metastatic disease | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics include those who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | GM-CSF Alone | pTVG-HP Vaccine With GM-CSF | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Median (Full Range); unit: years] | 71 [56 to 86] | 71 [46 to 82] | 71 [46 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 49 | 48 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 46 | 43 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 97
Prior Treatment [Count of Participants; unit: Participants]
  Prostatectomy | 34 | 41 | 75
  Primary Radiation Therapy | 20 | 12 | 32
  Adjuvant Radiation Therapy | 28 | 31 | 59
  Androgen Deprivation | 13 | 15 | 28
  Chemotherapy | 1 | 1 | 2
Gleason Score [Count of Participants; unit: Participants] — Gleason grade (1-5 were 1 is normal cells and 5 is the most high-grade cells) is assigned to the most predominant biopsy pattern and a second Gleason grade to the second most predominant pattern. For example: 3 + 4. The two grades will then be added together to determine the Gleason score. A Gleason Score of 6 is low grade, 7 is intermediate, and 8 - 10 is high grade cancer.
  Participants
    less than or equal to 7 | 34 | 32 | 66
    greater than 7 | 15 | 16 | 31
Baseline Prostate-Specific Antigen (PSA) [Count of Participants; unit: Participants]
  2.0 - 10.0 ng/mL | 42 | 40 | 82
  greater than 10 ng/mL | 7 | 8 | 15
Baseline PSA Doubling Time [Count of Participants; unit: Participants]
  less than 3 months | 10 | 11 | 21
  3-6 months | 22 | 21 | 43
  6-12 months | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: 2-year Metastasis-Free Survival Rate
Description: 2-year Metastasis-Free Survival (MFS) Rate with the development of metastases by conventional imaging used to define progression (as defined by RECIST 1.1 criteria). The 2-year MFS rate estimates which were obtained using the Kaplan-Meier analysis (taking into account censoring) using the intention-to-treat population.
Time Frame: 2 years
Measure: Number; unit: percent probability
Arm/Group | GM-CSF Alone | pTVG-HP Vaccine With GM-CSF
Number analyzed (Participants) | 49 | 48
percent probability | 42.3 | 41.8
Statistical Analysis 1: Comparison: GM-CSF Alone vs pTVG-HP Vaccine With GM-CSF; Test type: Other; p = 0.97, Mantel Haenszel

2. Secondary Outcome: Prostate Specific Antigen (PSA) Doubling Time (DT)
Description: PSA DT was calculated using all serum PSA values available from the same clinical laboratory for the specified period by the equation log2/b where b denotes the least-squares estimator of the linear regression model of the log-transformed PSA values on time. Pretreatment PSA DT (3-6 months before treatment, with a minimum of 4 values), on-treatment PSA DT was determined using values from month 3 to month 9.
Time Frame: up to 9 months
Measure: Median (Full Range); unit: months
Arm/Group | GM-CSF Alone | pTVG-HP Vaccine With GM-CSF
Number analyzed (Participants) | 49 | 48
months | 8.9 [1.6 to 77.9] | 5.4 [1.8 to 77.9]
Statistical Analysis 1: Comparison: GM-CSF Alone vs pTVG-HP Vaccine With GM-CSF; Test type: Superiority; p = .08, Wilcoxon Rank Sum test

3. Secondary Outcome: Number and Severity of Observed Toxicities
Description: Number of participants who experienced any adverse events greater than grade 1 that were determined to be at least possibly related to treatment, highest grade reported per participant for each adverse event (AE). All toxicities were graded using National Cancer Institute Common Terminology Criteria for Adverse Events (version 4). Higher grades indicate more severe toxicities.
Time Frame: 2 years
Population: Number of Severity of Adverse Events (AE) by grade complements the Adverse Events Section of this record.
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF Alone | pTVG-HP Vaccine With GM-CSF
Number analyzed (Participants) | 49 | 48
Participants
  Chills: Grade 2 | 2 | 1
  Chills: Grade 3 | 0 | 0
  Chills: Grade 4 | 0 | 0
  Chills: Did not experience this AE | 47 | 47
  Fatigue: Grade 2 | 2 | 1
  Fatigue: Grade 3 | 0 | 0
  Fatigue: Grade 4 | 0 | 0
  Fatigue: Did not experience this AE | 47 | 47
  Injection Site Reaction: Grade 2 | 2 | 2
  Injection Site Reaction: Grade 3 | 0 | 0
  Injection Site Reaction: Grade 4 | 0 | 0
  Injection Site Reaction: Did not experience this AE | 47 | 46
  Nausea: Grade 2 | 0 | 1
  Nausea: Grade 3 | 0 | 0
  Nausea: Grade 4 | 0 | 0
  Nausea: Did not experience this AE | 49 | 47
  Allergic Reaction: Grade 2 | 3 | 0
  Allergic Reaction: Grade 3 | 0 | 1
  Allergic Reaction: Grade 4 | 0 | 0
  Allergic Reaction: Did not experience this AE | 46 | 47
  Shingles: Grade 2 | 0 | 1
  Shingles: Grade 3 | 0 | 0
  Shingles: Grade 4 | 0 | 0
  Shingles: Did not experience this AE | 49 | 47
  Sinusitis: Grade 2 | 0 | 1
  Sinusitis: Grade 3 | 0 | 0
  Sinusitis: Grade 4 | 0 | 0
  Sinusitis: Did not experience this AE | 49 | 47
  Arthritis: Grade 2 | 2 | 0
  Arthritis: Grade 3 | 0 | 0
  Arthritis: Grade 4 | 0 | 0
  Arthritis: Did not experience this AE | 47 | 48
  Generalized Muscle Weakness: Grade 2 | 0 | 1
  Generalized Muscle Weakness: Grade 3 | 0 | 0
  Generalized Muscle Weakness: Grade 4 | 0 | 0
  Generalized Muscle Weakness: Did not experience this AE | 49 | 47
  Myalgia: Grade 2 | 0 | 1
  Myalgia: Grade 3 | 0 | 0
  Myalgia: Grade 4 | 0 | 0
  Myalgia: Did not experience this AE | 49 | 47
  Headache: Grade 2 | 1 | 1
  Headache: Grade 3 | 0 | 0
  Headache: Grade 4 | 0 | 0
  Headache: Did not experience this AE | 48 | 47
  Paresthesia: Grade 2 | 0 | 1
  Paresthesia: Grade 3 | 0 | 0
  Paresthesia: Grade 4 | 0 | 0
  Paresthesia: Did not experience this AE | 49 | 47
  Syncope: Grade 2 | 0 | 0
  Syncope: Grade 3 | 0 | 1
  Syncope: Grade 4 | 0 | 0
  Syncope: Did not experience this AE | 49 | 47
  Rash: Grade 2 | 0 | 1
  Rash: Grade 3 | 0 | 0
  Rash: Grade 4 | 0 | 0
  Rash: Did not experience this AE | 49 | 47
  Skin Swelling: Grade 2 | 0 | 1
  Skin Swelling: Grade 3 | 0 | 0
  Skin Swelling: Grade 4 | 0 | 0
  Skin Swelling: Did not experience this AE | 49 | 47
  Hot Flashes: Grade 2 | 0 | 1
  Hot Flashes: Grade 3 | 0 | 0
  Hot Flashes: Grade 4 | 0 | 0
  Hot Flashes: Did not experience this AE | 49 | 47
  Hypertension: Grade 2 | 1 | 1
  Hypertension: Grade 3 | 0 | 2
  Hypertension: Grade 4 | 0 | 0
  Hypertension: Did not experience this AE | 48 | 45
  Increased ALT: Grade 2 | 0 | 1
  Increased ALT: Grade 3 | 0 | 0
  Increased ALT: Grade 4 | 0 | 0
  Increased ALT: Did not experience this AE | 49 | 47
  Increased AST: Grade 2 | 0 | 1
  Increased AST: Grade 3 | 0 | 0
  Increased AST: Grade 4 | 0 | 0
  Increased AST: Did not experience this AE | 49 | 47
  Decreased ANC: Grade 2 | 0 | 0
  Decreased ANC: Grade 3 | 0 | 1
  Decreased ANC: Grade 4 | 0 | 1
  Decreased ANC: Did not experience this AE | 49 | 46
  Decreased WBC: Grade 2 | 0 | 1
  Decreased WBC: Grade 3 | 0 | 0
  Decreased WBC: Grade 4 | 0 | 0
  Decreased WBC: Did not experience this AE | 49 | 47

4. Secondary Outcome: Median Time to Radiographic Disease Progression
Description: Time to metastasis was determined from the date of registration to the first CT or bone scan that demonstrated metastatic disease. As defined by RECIST 1.1 criteria.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GM-CSF Alone | pTVG-HP Vaccine With GM-CSF
Number analyzed (Participants) | 49 | 48
months | 18.3 [12.3 to 24.2] | 18.9 [12.0 to 24.9]
Statistical Analysis 1: Comparison: GM-CSF Alone vs pTVG-HP Vaccine With GM-CSF; Test type: Other; p = 0.14, Regression, Cox; Hazard Ratio (HR) = 1.6, 95% CI 2-sided [0.9 to 2.8]

5. Secondary Outcome: PSA Progression Free Survival
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GM-CSF Alone | pTVG-HP Vaccine With GM-CSF
Number analyzed (Participants) | 49 | 48
months | 9.0 [8.8 to 12.0] | 8.9 [6.0 to 11.8]

ADVERSE EVENTS:
Time Frame: up to 2 years
Description: Adverse Events data for all participants who started the study.
Arm/Group | GM-CSF Alone | pTVG-HP Vaccine With GM-CSF
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 6/49 | 3/50
Other Adverse Events (participants affected / at risk) | 45/49 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GM-CSF Alone (N=49) | pTVG-HP Vaccine With GM-CSF (N=50)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac disorders (Cardiac disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nervous system disorders - other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GM-CSF Alone (N=49) | pTVG-HP Vaccine With GM-CSF (N=50)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 1 (4)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (3) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 2 (3)
Watering Eyes (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (5)
Anal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (13)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Chills (General disorders) | 6 (7) | 5 (12)
Edema limbs (General disorders) | 3 (3) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 17 (51) | 20 (38)
Fever (General disorders) | 4 (7) | 3 (3)
Flu like symptoms (General disorders) | 6 (14) | 8 (30)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 34 (119) | 28 (104)
Localized edema (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 5 (14) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (4)
Pain (General disorders) | 9 (10) | 10 (13)
Allergic reaction (Immune system disorders) | 2 (2) | 4 (4)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2) | 3 (4)
skin infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0)
Cholesterol high (Investigations) | 2 (2) | 0 (0)
Investigations - Other, specify (Investigations) | 3 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 1 (1)
Anorexia (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 3 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 10 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (11) | 6 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 7 (13) | 9 (17)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 11 (36) | 7 (14)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (2) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 3 (4)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2) | 5 (6)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0)
Nail Ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (9) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 2 (3)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 3 (8) | 2 (2)
Hypertension (Vascular disorders) | 9 (11) | 8 (9)
Hypotension (Vascular disorders) | 0 (0) | 2 (3)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT01341652/Prot_SAP_000.pdf